CLINICAL TRIAL: NCT04350112
Title: An Observational Study of Diagnostic Criteria, Clinical Features and Management of Opioid-induced Constipation (OIC) in Patients With Cancer Pain
Brief Title: Study of Opioid-Induced Constipation 1 Project
Acronym: StOIC-1
Status: Completed | Type: Observational
Sponsor: Royal Surrey County Hospital NHS Foundation Trust (Other)
Collaborators: Kyowa Hakko Kirin UK, Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: StOIC-1 Project
Record Dates: First submitted 2020-04-13; First posted 2020-04-16 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Opioid-induced Constipation; Cancer; Cancer Pain
Keywords: Opioid-induced constipation
MeSH Terms: conditions — Opioid-Induced Constipation; Neoplasms; Cancer Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Clinical assessment — Clinical assessment (history, examination) is gold standard for diagnosing constipation - gold standard will be compared with simple question about constipation, Rome IV diagnostic criteria for OIC, and common definitions of constipation for constipation / OIC

SUMMARY:
The aim of the project is to investigate opioid-induced constipation (OIC) in a real world / diverse group of patients with cancer.

The objectives of the project are to determine: a) prevalence of OIC; b) clinical features / impact of OIC; c) management of OIC.

DETAILED DESCRIPTION:
StOIC-1 is an observational study, and will involve a single visit (see below for schedule).

The following data will be collected: a) demographic data - age, gender, ethnicity; b) cancer diagnosis; c) opioid medications - drug, formulation, dose; d) laxative medications - drug, formulation, dose; e) other medications; f) Eastern Co-operative Oncology Group performance status

The participants will be asked the following questions:

1. Simple question - "Are you constipated?" [Options - yes / no / unsure]
2. European Association for Palliative Care definition question - "Does the following question describe your bowel function: 'the passage of small, hard faeces infrequently and with difficulty?' [Options - yes / no / unsure]
3. Camilleri definition question - "Does the following statement describe your bowel function: 'a change since initiating opioid therapy from baseline bowel habits that is characterised by any of the following: reduced bowel movement frequency, development or worsening of straining to pass bowel movements, a sense of incomplete rectal evacuation, harder stool consistency?' [Options - yes / no / unsure
4. Rome IV diagnostic criteria for OIC

The participants will also be asked to complete:

1. Bowel function index (BFI). The BFI is a validated, 3 item, patient-reported tool for assessing the treatment of OIC. A BFI score of ≥30 indicates suboptimally treated OIC.
2. Patient Assessment of Constipation - Quality of Life Questionnaire (PAC-QOL). The PAC-QOL is a validated, 28-item, patient-reported tool for assessing the impact of constipation over time.
3. Memorial Symptom Assessment Scale - Short Form (MSAS-SF). The MSAS-SF is a validated, 32 item, patient-reported tool for assessing physical and psychological symptoms in cancer patients.

The participant will also undergo a palliative care specialist assessment for constipation / OIC. The palliative care specialist will be asked to review the patient with regard to their bowel function, and then asked the following questions: a) does the patient have constipation? [Options - yes / no / unsure]; b) (if appropriate) does the patient have opioid-induced constipation? [Options - yes / no / unsure]; c) (if appropriate) does the patient have additional causes of constipation? [Options - yes / no / unsure]; d) (if appropriate) what additional causes of constipation?I

ELIGIBILITY:
Inclusion Criteria:

* Age > 18yr; diagnosis of cancer; diagnosis of cancer pain; receipt of regular opioids for at least one week

Exclusion Criteria:

* Inability to give informed consent; inability to complete questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1000 subjects that are either inpatients or outpatients at study sites (hospitals and hospices in the United Kingdom)
Sampling Method: Non-Probability Sample
Enrollment: 1007 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of opioid-induced constipation | 1 week
  Clinician assessment

CONTACTS AND LOCATIONS:
Overall Officials: Andrew N Davies, MD, Principal Investigator — Consultant Palliative Medicine
Locations (16):
- United Kingdom (16):
  - Royal Cornwall Hospital, Truro, Cornwall
  - Brighton & Sussex University Hospitals, Brighton, East Sussex
  - Leckhampton Court Hospice, Cheltenham, Gloucestershire
  - Hospice of St. Francis, Berkhamstead, Hertfordshire
  - Heart of Kent Hospice, Maidstone, Kent
  - Wisdom Hospice, Rochester, Kent
  - St. Raphael's Hospice, Cheam, London
  - Nottingham University Hospitals, Nottingham, Nottinghamshire
  - St Margaret's Hospice, Yeovil, Somerset
  - St. Giles Hospice, Lichfield, Staffordshire
  - Royal Surrey County Hospital, Guildford, Surrey
  - Birmingham St. Mary's Hospice, Birmingham, West Midlands
  - St. Catherine's Hospice, Crawley, West Sussex
  - St. Gemma's Hospice, Leeds, Yorkshire
  - Wheatfields Hospice, Leeds, Yorkshire
  - St. Luke's Hospice, Sheffield, Yorkshire

IPD SHARING:
Plan to Share IPD: No
Currently, there are no plans to make IPD available to other researchers

REFERENCES:
- [Result] Camilleri M, Drossman DA, Becker G, Webster LR, Davies AN, Mawe GM. Emerging treatments in neurogastroenterology: a multidisciplinary working group consensus statement on opioid-induced constipation. Neurogastroenterol Motil. 2014 Oct;26(10):1386-95. doi: 10.1111/nmo.12417. Epub 2014 Aug 28. PMID 25164154
- [Result] Larkin PJ, Sykes NP, Centeno C, Ellershaw JE, Elsner F, Eugene B, Gootjes JR, Nabal M, Noguera A, Ripamonti C, Zucco F, Zuurmond WW; European Consensus Group on Constipation in Palliative Care. The management of constipation in palliative care: clinical practice recommendations. Palliat Med. 2008 Oct;22(7):796-807. doi: 10.1177/0269216308096908. PMID 18838491
- [Result] Mearin F, Lacy BE, Chang L, Chey WD, Lembo AJ, Simren M, Spiller R. Bowel Disorders. Gastroenterology. 2016 Feb 18:S0016-5085(16)00222-5. doi: 10.1053/j.gastro.2016.02.031. Online ahead of print. PMID 27144627
- [Result] Argoff CE, Brennan MJ, Camilleri M, Davies A, Fudin J, Galluzzi KE, Gudin J, Lembo A, Stanos SP, Webster LR. Consensus Recommendations on Initiating Prescription Therapies for Opioid-Induced Constipation. Pain Med. 2015 Dec;16(12):2324-37. doi: 10.1111/pme.12937. Epub 2015 Nov 19. PMID 26582720
- [Result] Chang VT, Hwang SS, Feuerman M, Kasimis BS, Thaler HT. The memorial symptom assessment scale short form (MSAS-SF). Cancer. 2000 Sep 1;89(5):1162-71. doi: 10.1002/1097-0142(20000901)89:53.0.co;2-y. PMID 10964347
- [Result] Marquis P, De La Loge C, Dubois D, McDermott A, Chassany O. Development and validation of the Patient Assessment of Constipation Quality of Life questionnaire. Scand J Gastroenterol. 2005 May;40(5):540-51. doi: 10.1080/00365520510012208. PMID 16036506
- [Result] Rentz AM, Yu R, Muller-Lissner S, Leyendecker P. Validation of the Bowel Function Index to detect clinically meaningful changes in opioid-induced constipation. J Med Econ. 2009;12(4):371-83. doi: 10.3111/13696990903430481. PMID 19912069
- [Result] Ueberall MA, Muller-Lissner S, Buschmann-Kramm C, Bosse B. The Bowel Function Index for evaluating constipation in pain patients: definition of a reference range for a non-constipated population of pain patients. J Int Med Res. 2011;39(1):41-50. doi: 10.1177/147323001103900106. PMID 21672306